CLINICAL TRIAL: NCT04855110
Title: Early Versus Late Post Caesarean Section Oral Anticoagulation Initiation and Risk of Maternal Complications in Patients With Mechanical Heart Valve Prosthesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Samir Fouad, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD-201-2020
Record Dates: First submitted 2021-04-19; First posted 2021-04-22 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Maternal Complications After Oral Anticoagulation When Initiated Early and Late After Caesarean Section Done for Patients With Mechanical Heart Valve Prosthesis
Keywords: oral anticoagulants, mechanical heart valve prosthesis, caesarean section, maternal complications

STUDY DESIGN:
Intervention Model Description: 114 pregnant women with mechanical prosthetic mitral and/or aortic valves, will be divided equally into 2 groups.Using a table of random numbers, participants will be divided into 2 equal groups. Group A (57 patients) in which warfarin will be started day 2 after caesarean delivery (i.e. 24 hours postoperative), and group B (57 patients) in which warfarin will be started day 5 after caesarean delivery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Day 2 warfarin group (Active Comparator): warfarin will be administered on day 2 after caesarean section (in a dose that achieves therapeutic level as indicated by the cardiology consultant)
  Interventions: Drug: Warfarin Sodium started on Day 2 after caesarean section (in a dose that achieves a therapeutic level as indicated by the cardiology consultant)
- Day 5 warfarin group (Active Comparator): warfarin will be administered on day 5 after caesarean section (in a dose that achieves therapeutic level as indicated by the cardiology consultant)
  Interventions: Drug: Warfarin Sodium started on day 5 after caesarean section (in a dose that achieves a therapeutic level as indicated by the cardiology consultant)

INTERVENTIONS:
Drug: Warfarin Sodium started on Day 2 after caesarean section (in a dose that achieves a therapeutic level as indicated by the cardiology consultant) — Warfarin started on day 2 after caesarean section in patients with mechanical heart valve prosthesis
  Arms: Day 2 warfarin group
Drug: Warfarin Sodium started on day 5 after caesarean section (in a dose that achieves a therapeutic level as indicated by the cardiology consultant) — Warfarin started on day 5 after caesarean section in patients with mechanical heart valve prosthesis
  Arms: Day 5 warfarin group

SUMMARY:
A randomized cohort study applied to patients with mechanical heart valve prosthesis who will be delivered by caesarean section at or after 28 weeks of gestation . Using a table of random numbers, participants will be divided into 2 equal groups. Group A (57 patients) in which warfarin will be started day 2 after caesarean delivery (i.e. 24 hours postoperative), and group B (57 patients) in which warfarin will be started day 5 after caesarean delivery, then maternal complications are compared among these 2 groups.

DETAILED DESCRIPTION:
-Background and Rationale:

Cardiac valve replacement surgery has saved the lives of hundreds of thousands of patients with acquired (e.g. rheumatic) or congenital cardiac disorders (McLintock, 2011).

Pregnancy induces a state of hypercoagulability with a high risk of thromboembolism. The thromboembolic risks are much higher in patients with mechanical prosthetic heart valves (Hanania, 2001).

Vitamin K antagonists (VKAs) constitute the safest anticoagulation for mechanical heart valves (MHV) whether within or outside of pregnancy. However, these drugs can cross the placenta and can cause embryopathy, fetopathy, and bleeding. In the peripartum period, there is also an increase in the bleeding risk for both, the mother and the neonate. (Bhagra et al, 2017).

On the other hand, heparins, both unfractionated (UFH) and low molecular weight heparin (LMWH), do not cross the placenta and are considered safe for the fetus. However, heparin seems an inadequate anticoagulant when used for MHV over long periods such as in pregnancy. This is due in part to the thrombogenic nature of MHV (Arya, 2019).

The preferred approach from the European society of cardiology (ESC) is the sequential use of heparin (LMWH or UFH) in the first trimester, VKAs in second and third trimesters reverting to heparin at 36 weeks gestation. If the warfarin dose required to reach the therapeutic international normalized ratio (INR) is 5 mg or less, it is suggested that warfarin could be continued in the first trimester. Therapeutic heparin (either unfractionated or low molecular weight) should be restarted 4-6 hours after delivery as long as the patient has no significant bleeding, then oral anticoagulants (VKAs) are introduced together with heparin till INR reaches the therapeutic level (Regitz-Zagrosek et al,2019).

After delivery, patients with mechanical heart valves are at significant risk of maternal morbidity and mortality. Morbidity includes primary and secondary postpartum hemorrhage, wound hematoma, intra-abdominal bleeding, need for reopera¬tion or other intervention, valve thrombosis, and other thromboembolic manifestations e.g. Stroke. However, there is limited guidance on when to start oral anticoagulants in the postpartum period (Irani et al, 2018).

Pooled institutional data and an interdisciplinary approach are recommended to minimize competing risks, sequelae of valve thrombosis, and obstetrical hemorrhage and, thereby, to optimize maternal outcomes and develop evidence-based guidelines for postpartum anticoagulation management (Irani et al, 2018).

Based on our observations at the high-risk pregnancy department in Kasr Al Ainy school of medicine, we noticed that the postpartum bleeding complications were different when oral anticoagulants (VKAs) were started on different days after cesarean section as we found that postpartum bleeding was noticeably less when warfarin was started 5 days after cesarean section, so we decided to conduct this study to address the appropriate timing to start oral anticoagulants after cesarean section.

-Population of study:

Pregnant women presenting to Kasr Al Ainy high risk pregnancy outpatient clinic with mechanical prosthetic mitral and/or aortic valves, and indicated to deliver via caesarean section at or after 28 weeks of gestation.

- Study location: Study will be conducted in Kasr Al Ainy high risk pregnancy unit. Participants will be recruited from Kasr Al Ainy high risk pregnancy outpatient clinic.

* Inclusion criteria:

  • Pregnant women with mechanical prosthetic heart valves who are planned to deliver by caesarean delivery, provided that the gestational age at delivery is 28 weeks of gestation or more whether singleton or multi-fetal pregnancy.
* Exclusion criteria:

  * Patients with right sided mechanical heart valves.
  * Patients with history of any thrombotic events e.g. Stuck prosthetic valve, or cerebrovascular stroke, etc.
  * Patients with hypertensive disorders.
  * Diabetic patients.
  * Patients with known bleeding disorders or coagulation defects.
  * Patients with known thrombophilia.
  * Patients who refuse to share in the study.
* Methodology in details:

A randomised (using tables of random numbers for randomization), cohort study, including 114 pregnant women presenting to Kasr Al Ainy high risk pregnancy outpatient clinic with mechanical prosthetic mitral and/or aortic valves.

After taking a written consent from all participants, they will be subjected to thorough history taking regarding age, parity, gestational age on presentation, medical history, duration since cardiac surgery, type and number of replaced valves, average dose of warfarin used during pregnancy, type and dose of anticoagulant immediately used before delivery, history of prosthetic valve complications and history of obstetric complications. General examination including maternal weight and height and abdominal (obstetric) examination will be performed. Antenatal ultrasonography will be done to determine gestational age and to assess for fetal wellbeing, then all patients will be examined by a Cardiology consultant to assess the cardiac status, adjust the anticoagulation dose, follow up for the occurrence of any cardiac complications, and to help in determining when to terminate and mode of termination according to individual patient's situation.

Starting from 36 weeks of gestation, all patients will be reverted to unfractionated heparin in a therapeutic dose (as determined by the cardiology consultant) to maintain activated partial thromboplastin time (aPTT) within a therapeutic level. Unfractionated heparin will be stopped 6 hours before caesarean section.

Participants who will be indicated to deliver via caesarean section (upon obstetric or cardiac recommendations), will be included, and will be operated upon by the same surgical team.

Routine preoperative labs including complete blood count, coagulation profile (to ensure that the PC is >60% and the INR is <1.5 prior to surgery), liver and kidney functions, and fasting and 2 hours postprandial blood sugar level will be withdrawn.

During caesarean section, adequate hemostasis will be achieved, an intraperitoneal drain will be inserted, parietal peritoneum will be closed, gel foams, and suction drain in the sub-rectus space will be inserted. After delivery, heparin will be started 4-6 hours and then switched to low molecular weight heparin (LMWHs) 12 hours after caesarean section, in the absence of significant bleeding, in twice daily subcutaneous injections in a therapeutic dose (1 mg/kg twice daily) (James 2011).

Using a table of random numbers, participants will be divided into 2 equal groups. Group A (57 patients) in which warfarin will be started day 2 after caesarean delivery (i.e. 24 hours postoperative), and group B (57 patients) in which warfarin will be started day 5 after caesarean delivery. In both groups, LMW heparin will be continued in a therapeutic dose as mentioned above beside warfarin till INR achieves a therapeutic value as determined by the cardiologist. When a therapeutic level of warfarin is achieved, LMW heparin will be stopped, patient will continue on warfarin, and will be discharged from the hospital. Duration till control of the INR will be reported in both groups.

For all participants, the amount of blood in the sub-rectus and intraperitoneal drains will be recorded. Clinical examination as well as transabdominal ultrasonography will be performed daily till the end of hospital stay, then 1 and 2 weeks after delivery to check for signs of wound hematoma . The ultrasonographic findings suggesting the presence of subcutaneous or sub-rectus hematoma include; a homogeneous or heterogeneous fluid collection within the abdominal wall, and Doppler colour flow which does not reliably detect the presence of active extravasation, then the size of hematoma will be measured in centimetres, and will be followed up in the daily consecutive ultrasonography examinations (Allen and Sevensma 2019).

For all patients, Other maternal outcomes will be recorded including primary postpartum hemorrhage, intra-abdominal bleeding, need for blood transfusion, need for reoperation e.g. re-exploration in case of significant intraperitoneal hemorrhage or evacuation of wound hematoma, or other intervention ( e.g. re-do cardiac valve replacement surgery in cases with stuck valve), valve thrombosis, other thromboembolic manifestations e.g. stroke, length of hospital stay, and maternal death. The timing and indication for caesarean delivery will be identified.

Postoperative haemoglobin and haematocrit values will be done 24 hours after the end of the operation as well as at the end of hospital stay before discharge. Estimation of intraoperative blood loss will be obtained through measuring the volume of blood in the suction machine reservoir and weighing the swabs (surgical towels) as soon as possible. The weights of dry swabs will be subtracted from the weights of swabs used during the operation. The weight of swabs found in grams will be translated to ml by using blood density (1.050 g/ml) (Caglar et al 2008).

Postoperative blood loss in the first 24 hours and after will be measured by subtracting intraoperative blood loss from total blood loss.

Total blood loss will be measured through pre and postoperative hematocrit values through the following equations:

The estimated total blood loss will be derived by multiplying the calculated pregnancy blood volume by percentage of blood volume lost.

* Pregnancy blood volume = (0.75 × {[maternal height (inches) × 50] + [maternal weight in pounds × 25]})
* Percent of blood volume lost = ({predelivery HCT - postdelivery HCT}/predelivery HCT)
* Total blood loss = pregnancy blood volume × percent of blood volume lost (Stafford et al, 2008)

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with mechanical prosthetic heart valves who are planned to deliver by caesarean delivery, provided that the gestational age at delivery is 28 weeks of gestation or more whether singleton or multi-fetal pregnancy.

Exclusion Criteria:

* Patients with right-sided mechanical heart valves.
* Patients with a history of any thrombotic events e.g. Stuck prosthetic valve, or cerebrovascular stroke, etc.
* Patients with hypertensive disorders.
* Diabetic patients.
* Patients with known bleeding disorders or coagulation defects.
* Patients with known thrombophilia.
* Patients who refuse to share in the study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — female pregnant women with a mechanical heart valve prosthesis
Enrollment: 114 (Estimated)
Dates: Start 2021-04-19 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Occurrence of subcutaneous and / or sub-rectus hematoma | 14 days
Occurrence of intra-abdominal bleeding | 14 days
Need for blood transfusion | 14 days
Need for abdominal re-exploration or wound hematoma evacuation | 14 days
Need for any other intervention e.g. redo valve replacement surgery in case of a stuck valve | 14 days
Occurrence of a valve thrombosis or other thromboembolic manifestations e.g. stroke | 14 days
Maternal death | 14 days

SECONDARY OUTCOMES:
Estimation of the average total intraoperative and postoperative blood loss in the first 24 hours after caesarean section | 24 hours
Length of hospital stay since delivery till discharge | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Maged A Abdel Raouf, professor, Study Director — Cairo University
Locations (1):
- Faculty of medicine (Kasr Alainy), cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arya R. Pregnancy outcomes in women with mechanical prosthetic heart valves. Thromb Res. 2019 Sep;181 Suppl 1:S37-S40. doi: 10.1016/S0049-3848(19)30365-2. PMID 31477226
- [Background] Bhagra CJ, D'Souza R, Silversides CK. Valvular heart disease and pregnancy part II: management of prosthetic valves. Heart. 2017 Feb;103(3):244-252. doi: 10.1136/heartjnl-2015-308199. Epub 2016 Sep 26. No abstract available. PMID 27670966
- [Background] Caglar GS, Tasci Y, Kayikcioglu F, Haberal A. Intravenous tranexamic acid use in myomectomy: a prospective randomized double-blind placebo controlled study. Eur J Obstet Gynecol Reprod Biol. 2008 Apr;137(2):227-31. doi: 10.1016/j.ejogrb.2007.04.003. Epub 2007 May 11. PMID 17499419
- [Background] Hanania G. Management of anticoagulants during pregnancy. Heart. 2001 Aug;86(2):125-6. doi: 10.1136/heart.86.2.125. No abstract available. PMID 11454818
- [Background] Irani RA, Santa-Ines A, Elder RW, Lipkind HS, Paidas MJ, Campbell KH. Postpartum anticoagulation in women with mechanical heart valves. Int J Womens Health. 2018 Oct 25;10:663-670. doi: 10.2147/IJWH.S177547. eCollection 2018. PMID 30498374
- [Background] Practice bulletin no. 123: thromboembolism in pregnancy. Obstet Gynecol. 2011 Sep;118(3):718-729. doi: 10.1097/AOG.0b013e3182310c4c. PMID 21860313
- [Background] McLintock C. Anticoagulant therapy in pregnant women with mechanical prosthetic heart valves: no easy option. Thromb Res. 2011 Feb;127 Suppl 3:S56-60. doi: 10.1016/S0049-3848(11)70016-0. PMID 21262443
- [Background] Regitz-Zagrosek V, Roos-Hesselink JW, Bauersachs J, Blomstrom-Lundqvist C, Cifkova R, De Bonis M, Iung B, Johnson MR, Kintscher U, Kranke P, Lang IM, Morais J, Pieper PG, Presbitero P, Price S, Rosano GMC, Seeland U, Simoncini T, Swan L, Warnes CA. 2018 ESC Guidelines for the management of cardiovascular diseases during pregnancy. Kardiol Pol. 2019;77(3):245-326. doi: 10.5603/KP.2019.0049. No abstract available. PMID 30912108
- [Background] Stafford I, Dildy GA, Clark SL, Belfort MA. Visually estimated and calculated blood loss in vaginal and cesarean delivery. Am J Obstet Gynecol. 2008 Nov;199(5):519.e1-7. doi: 10.1016/j.ajog.2008.04.049. Epub 2008 Jul 17. PMID 18639209
- [Background] van Hagen IM, Roos-Hesselink JW, Ruys TP, Merz WM, Goland S, Gabriel H, Lelonek M, Trojnarska O, Al Mahmeed WA, Balint HO, Ashour Z, Baumgartner H, Boersma E, Johnson MR, Hall R; ROPAC Investigators and the EURObservational Research Programme (EORP) Team*. Pregnancy in Women With a Mechanical Heart Valve: Data of the European Society of Cardiology Registry of Pregnancy and Cardiac Disease (ROPAC). Circulation. 2015 Jul 14;132(2):132-42. doi: 10.1161/CIRCULATIONAHA.115.015242. Epub 2015 Jun 22. PMID 26100109
- [Derived] Youssef G, Mohamed TEH, Abdel Raouf MA, Fouad Tammam AS, Gabr AA. Early Versus Late Post Cesarean Section Warfarin Initiation and Increased Risk of Maternal Complications in Patients With Mechanical Heart Valves: A Randomized, Open-Label Pilot Study. Korean Circ J. 2025 Feb;55(2):151-160. doi: 10.4070/kcj.2024.0002. Epub 2024 Jul 3. PMID 39175342